CLINICAL TRIAL: NCT04505059
Title: Effect of Different Anesthetic Strategies on Postoperative Cognitive Function and Delirium in Adult Patients Undergoing Cardiac Surgery
Brief Title: Different Anesthetic Strategies on Postoperative Cognitive Function and Delirium in Patients Undergoing Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Tianjin Chest Hospital (Other); The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Yuefu Wang, Professor, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Precision-Delirium-Cognitive
Record Dates: First submitted 2020-07-18; First posted 2020-08-07 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-01

CONDITIONS: Delirium; Condition; Anesthesia
Keywords: Postoperative cognitive function; Delirium; Cardiac Surgical Procedures; Precision cardiac anesthesia
MeSH Terms: conditions — Delirium; Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precision cardiac anesthesia (Experimental): Remifentanil (TCI) for intra-operative analgesia Propofol (TCI) for intra-operative sedation
  Interventions: Procedure: Precision cardiac anesthesia
- Conventional cardiac anesthesia (Active Comparator): Institutional standard of care.
  Interventions: Procedure: Conventional cardiac anesthesia

INTERVENTIONS:
Procedure: Precision cardiac anesthesia — Aperi-operative anesthetic management through target-controlled infusion to accurately control the patient blood concentration, with combination of bispectral index and neuromuscular monitoring to adjust the dosage of general anesthetics.
  Arms: Precision cardiac anesthesia
Procedure: Conventional cardiac anesthesia — The anesthesia strategy is mainly depending on the anesthesiologist's clinical experience
  Arms: Conventional cardiac anesthesia

SUMMARY:
This is a prospective, multi-center, double-blind, randomized clinical trials.

DETAILED DESCRIPTION:
Prospective randomized multi-center trial involving about 502 subjects will be enrolled in 3 centers. Patients will be randomized to two groups in equal proportion. Investigators set a hypothesis that precision cardiac anesthesia, which involves the modification of several crucial anesthetic modalities, would reduces the incidence of postoperative cognitive function and delirium in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged≥18 years;
2. ASA:I to III;
3. Hemodynamic stability, LVEF≥40%;
4. Cardiac surgery including CABG, valve surgery, CABG combined with valve surgery, surgical repair of ASD,VSD and atrial myxoma, and other types.

Exclusion Criteria:

1. Declined to get involved;
2. Emergency cases, heart transplantation;
3. Severe hepatic insufficiency (Child-Pugh grades C),Severe renal insufficiency (requirement of renal replacement therapy);
4. Previous history of drug and alcohol abuse,allergy to general anesthetics;
5. Preoperative severe dementia, language barrier and mental illness
6. Preoperative schizophrenia, epilepsy, stroke and Parkinson's disease
7. Previous history of craniocerebral injury or neurosurgery;
8. Any other conditions that are considered unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2022-07-18 (Estimated); Study Completion 2023-01-18 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperative delirium | Postoperative day 1 to 5
  Delirium assessed by using Confusion Assessment Method-ICU (CAM-ICU) in the postoperative period

SECONDARY OUTCOMES:
Postoperative cognitive function | In hospital,up to 10 days, at 1,6 and 12 months after surgery
  Assessed by MoCA (score range from 0 to 30, higher scores mean a better outcome) or MMSE (score range from 0 to 30, higher scores mean a better outcome)
Ventilation time | up to 1 month after surgery
  Mechanical ventilation time after surgery
Length of stay | up to 2 months after surgery
  Length of hospital and ICU stay
Cost | up to 2 months after surgery
  health care costs of hospital and ICU
PONV | Postoperative day 1 to 5
  To quantify postoperative nausea and vomiting the following score was used:
  0 = no nausea, 1 = nausea, 2 = retching, 3 = single vomiting, 4 = multiple vomiting.
Postoperative pain | Postoperative day 1 to 5, at 1,6 and 12 months after surgery
  Assessed by NRS (from 0 to 10, higher scores mean a worse outcome)
IL-6, IL-8, IL-10 | Before surgery, 6h, postoperative day 1 (POD1) morning, 24h,after surgery
  Inflammatory factor (IL-6, IL-8, IL-10)
TNF-α | Before surgery, 6h, postoperative day 1(POD1 )morning, 24h after surgery
  Inflammatory factor (TNF-α)
IGF-1 | Before surgery, 6h, postoperative day 1 (POD1) morning, 24h after surgery
  Blood Biomarker (IGF-1)
CRP | Before surgery, 6h, postoperative day 1 (POD1) morning, 24h after surgery
  Blood Biomarker (CRP)
S-100β protein | Before surgery, 6h, postoperative day 1 (POD1) morning, 24h after surgery
  Blood Biomarker (S-100β protein)
Genotype | Before surgery
  Number of participants with target gene

OTHER OUTCOMES:
Rate of postoperative complications | In hospital,up to 10 days, at 1,3 and 12 months after surgery
  Postoperative main complications
Rate of mortality | In hospital,up to 10 days, at 1,3 and 12 months after surgery
  All-cause mortality
Patient's life quality | At 1,3 and 12 months after surgery
  Quality of life was assessed by SF-36. A self-administered 36-item question- naire covering eight different domains: physical functioning, physical role functioning, bodily pain, general health, vitality, social functioning, emotional role functioning, and mental health. Raw points are transformed into a score from 0 to 100 for each dimension, with 100 reflecting the best possible health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yuefu Wang, MD, Study Director — Fuwai Hospital, China National Center for Cardiovascular Diseases, CAMS&PUMC; Jiange Han, MD, Principal Investigator — Tianjin Chest Hospital; Haitao Liu, MD, Principal Investigator — The Second Hospital of Hebei Medical University
Locations (3):
- China (3):
  - The Second Hospital of HeBei Medical University, Shijiazhuang, Hebei
  - Fuwai Hospital, China National Center for Cardiovascular Diseases, CAMS&PUMC, Beijing
  - Tianjin Chest Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No